CLINICAL TRIAL: NCT01603264
Title: Phase 1, Double Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Comparative Pharmacokinetic Study Of PF-05280014 And Trastuzumab Sourced From US And EU Administered To Healthy Male Volunteers
Brief Title: A Pharmacokinetic Study Comparing PF-05280014 And Trastuzumab In Healthy Male Volunteers (REFLECTIONS B327-01)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B3271001; REFLECTIONS B327-01
Record Dates: First submitted 2012-05-14; First posted 2012-05-22 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Bioequivalence; Biosimilarity; Similarity; PK; Phase I; Trastuzumab; Healthy Male Volunteers; Single-dose; HER-2; Oncology
MeSH Terms: conditions — Neoplasms | interventions — PF-05280014; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): PF-05280014
  Interventions: Biological: PF-05280014
- B (Active Comparator): Trastuzumab-EU
  Interventions: Biological: Herceptin
- C (Active Comparator): Trastuzumab-US
  Interventions: Biological: Herceptin

INTERVENTIONS:
Biological: PF-05280014 — Concentrate for solution for infusion, sterile vial 150 mg, single-dose 6 mg/kg administered as 90-minute infusion on day 1
  Other Names: Trastuzumab-Pfizer
  Arms: A
Biological: Herceptin — Concentrate for solution for infusion, sterile vial 150 mg, single-dose 6 mg/kg administered as 90-minute infusion on day 1
  Other Names: Trastuzumabum (European Union)
  Arms: B
Biological: Herceptin — Concentrate for solution for infusion, sterile vial 440 mg, single-dose 6 mg/kg administered as 90-minute infusion on day 1
  Other Names: Trastuzumab (United States)
  Arms: C

SUMMARY:
In this study, healthy male volunteers will receive a single intravenous administration of either PF-05280014 or trastuzumab (United States) or trastuzumab (European Union). During the course of the study, the pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms of PF-05280014 and the US-licensed and EU-approved trastuzumab products. Safety, tolerability, and immunologic response also will be evaluated throughout.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects (healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination including blood pressure and pulse rate measurement, 12-lead ECG, and clinical laboratory tests). Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight > 50 kg (110 lbs).
* Male subjects must agree that they and their female spouse/partners will use adequate contraception (2 forms of birth control, one of which must be barrier method) or be of non-childbearing potential.
* Left ventricular ejection fraction (LVEF) within the normal range as measured by echocardiogram (ECHO) within 8 weeks prior to randomization.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic or allergic disease, or clinical findings at screening excluding untreated, asymptomatic seasonal allergies at time of dosing.
* Clinically significant abnormalities in laboratory test results.
* Previous exposure to a monoclonal antibody or current use of other biologics.
* History of allergic or anaphylactic reaction to a therapeutic drug or benzyl alcohol.
* Use of prescription or non prescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements must be discontinued 28 days prior to the first dose of study medication.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters Area-Under-the-Curve (AUC) and Maximal Concentration (Cmax) of PF-05280014 compared to trastuzumab-EU. | Day 1 - Day 71
Pharmacokinetic parameters Area-Under-the-Curve (AUC) and Maximal Concentration (Cmax) of PF-05280014 compared to trastuzumab-US. | Day 1 - Day 71
Pharmacokinetic parameters Area-Under-the-Curve (AUC) and Maximal Concentration (Cmax) of trastuzumab-EU to trastuzumab-US. | Day 1 - Day 71

SECONDARY OUTCOMES:
Incidence of anti-trastuzumab antibodies (ADAs), including neutralizing antibodies (Nab). | Day 1 - LSLV or Day 71 whichever occurs later
Pharmacokinetic parameters Maximal Concentration (Cmax) and Area-Under-the-Curve (AUC) for the combined groups of trastuzumab-US and trastuzumab EU. | Day 1 - Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Yin D, Barker KB, Li R, Meng X, Reich SD, Ricart AD, Rudin D, Taylor CT, Zacharchuk CM, Hansson AG. A randomized phase 1 pharmacokinetic trial comparing the potential biosimilar PF-05280014 with trastuzumab in healthy volunteers (REFLECTIONS B327-01). Br J Clin Pharmacol. 2014 Dec;78(6):1281-90. doi: 10.1111/bcp.12464. PMID 25041377
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3271001&StudyName=A%20Pharmacokinetic%20Study%20Comparing%20PF-05280014%20And%20Trastuzumab%20In%20Healthy%20Male%20Volunteers%20%28REFLECTIONS%20B327-01%29